CLINICAL TRIAL: NCT04898881
Title: Breast Milk vs 24 % Sucrose in Procedural Pain Relief in Preterm Infants: Randomized Controlled Trial
Brief Title: Breast Milk vs Sucrose in Relieving Procedural Pain in Preterm Neonates During Blood Draw by Automated Heel Lance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Pradeep Velumula, Fellow, Neonatal-Perinatal Medicine, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1905002251
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Pain
Keywords: Pain management in preterm neonates
MeSH Terms: conditions — Pain | interventions — Milk, Human; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breast Milk (Active Comparator): 2 ml of Breast milk given one time, two minutes prior to the heel lance
  Interventions: Other: Breast Human Milk
- 24 %Sucrose (Other): 0.5 ml sucrose to be given once, two minutes prior to the heel lance
  Interventions: Other: 24 % Sucrose

INTERVENTIONS:
Other: Breast Human Milk — Interventional drug is given to the neonates 2 minutes before the heel lance
  Arms: Breast Milk
Other: 24 % Sucrose — 0.5 ml of sucrose given once 2 minutes prior to procedure
  Arms: 24 %Sucrose

SUMMARY:
Skin breaking procedure through an automated heel lancet for blood draws is a common painful procedure in the Neonatal Intensive care unit (NICU). Recurrent pain in preterm neonates is associated with long-term complications. The primary objective of the study is to compare pain scores between two groups (24% sucrose and breast milk) during blood draw using an automated heel lancet in preterm neonates. The investigator conducted a prospective randomized controlled trial in preterm neonates, to compare the pain scores in infants receiving either breast milk or sucrose. Premature Infant pain profile- Revised pain profile is used to assign pain scores. The primary outcome measure is the comparison of pain scores between the two groups.

DETAILED DESCRIPTION:
Blood draw by automated heel lancet is a common painful procedure in the Neonatal Intensive care units (NICU). The cutaneous sensory receptors on all mucosal and cutaneous surfaces are developed by 20 weeks gestational age (GA) and the neuronal circuits that carry pain stimuli from skin to cerebral cortex are developed by around 26 weeks of GA. Recurrent pain in preterm neonates impacts their postnatal growth, development, is associated with altered pain perception, and increased behavioral responses for future painful procedures.

Oral sucrose is a commonly administered and effective non-pharmacologic intervention used in the NICU for pain relief. There is insufficient evidence on its mechanism of action, minimum effective dose, the effect of repeated doses on long-term neurodevelopmental outcomes, and the consistency in providing pain relief with repeated doses over time. Moreover, the analgesic effect of sucrose is a developmentally transient phenomenon. Another non-pharmacologic intervention studied for pain relief in neonates is breast milk. The analgesic property of breast milk is presumed to be from its sweet taste from lactose, flavor, and odor. Breast milk has high levels of tryptophan, a melatonin precursor which may increase secretion of beta-endorphin, an endogenous opioid.

There is a paucity of data comparing analgesic properties of breast milk and sucrose in preterm neonates, along with insufficient evidence of sucrose as mentioned earlier, The investigator conducted this prospective randomized controlled trial (RCT) comparing sucrose with breast milk for pain relief in preterm neonates.

The primary objective of the study is to compare pain scores between two groups (24% sucrose and breast milk) during blood draw by automated heel lancet, in preterm neonates. The pain scores between the two groups will also be compared at 30 seconds intervals until two minutes post-procedure.

The current study is conducted at Hutzel Women's Hospital and Children's Hospital of Michigan NICU. Institutional Review Board approval was obtained from Wayne State University prior to study initiation. Before the study was initiated, physicians were trained in assessing the PIPP-R pain scale. The pain scores were given by two physicians who were blinded to the treatment arm, at baseline, during, 30-, 60-, 90-, and 120 seconds post-procedure. These scores were given either at the time of the procedure or a video is recorded to be scored later.

Eligible participants were identified and written informed consent was obtained from the parents. The timing and need for a blood draw are decided by the clinical team and are performed by the nurse taking care of the participant. Randomization was done by the pharmacist through a computer-generated program. Participants were randomly assigned to receive either 0.5 ml 24 % sucrose or 2 ml breastmilk, 2 minutes prior to the procedure. On the day of the procedure, the pharmacist sent a closed sealed envelope with a randomization group to the nurse taking care of the participant. Pain scores are given by two physicians during and post-procedure.

Te Investigators collected maternal characteristics of participants like age, prenatal care, race, history of diabetes and hypertension, receipt of antenatal steroids, magnesium, histological diagnosis of chorioamnionitis, mode of delivery, and duration of rupture of membranes. Neonatal characteristics collected include sex, APGAR score at 1 and 5 minutes, birth weight, gestational age, weight on the day of the procedure, postmenstrual age, number of skin pricks prior to the day of the procedure, and adverse events pre-defined as heart rate >240beats/minute or heart rate <80 beats/minute for >20 seconds, oxygen saturation <80 for >20 seconds, no spontaneous respiration for >20 seconds, choking, gagging were collected.

For this non-inferiority trial, the investigators chose the clinically significant difference to be 2 between the median PIPP-R scores during the procedure The investigators required 88 patients (44 in each group) to show that the lower limit of one-sided 95 % CI will be above the non-inferiority limit of -2 for an alpha error of 5% and power of 90 %.

ELIGIBILITY:
Inclusion Criteria:

1. All Infants with gestational age between 30 1/7 and 36 6/7 weeks
2. Within 30 days of post-natal life
3. Breast milk is available for the neonate
4. Scheduled for a blood draw

Exclusion Criteria:

1. Neonates on intravenous or peroral medications for sedation/analgesia or anti-epileptics
2. Infants diagnosed with neonatal abstinence syndrome and neonatal encephalopathy
3. Infants who are critically ill, on assisted ventilation > 2L HFNC and on ionotropic support
4. Infants with major congenital abnormalities/dysmorphism

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Pain Profile | During the Procedure
  Premature Infant Pain Profile- Revised pain profile is used to give pain scores to the participants. Minimum score and maximum scores on the scale are zero and twenty one. The pain scores increases with increasing severity of pain.

SECONDARY OUTCOMES:
Pain Profile | Pain scores will be given at 30 seconds interval for 2 minutes, post-procedure
  Premature Infant Pain Profile- Revised pain profile is used to give pain scores to the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Velumula, MD, Principal Investigator — Detroit Medical Center
Locations (1):
- Detroit Medical center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sener Taplak A, Erdem E. A Comparison of Breast Milk and Sucrose in Reducing Neonatal Pain During Eye Exam for Retinopathy of Prematurity. Breastfeed Med. 2017 Jun;12:305-310. doi: 10.1089/bfm.2016.0122. Epub 2017 Apr 17. PMID 28414522
- [Background] Shah PS, Herbozo C, Aliwalas LL, Shah VS. Breastfeeding or breast milk for procedural pain in neonates. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD004950. doi: 10.1002/14651858.CD004950.pub3. PMID 23235618
- [Background] Simonse E, Mulder PG, van Beek RH. Analgesic effect of breast milk versus sucrose for analgesia during heel lance in late preterm infants. Pediatrics. 2012 Apr;129(4):657-63. doi: 10.1542/peds.2011-2173. Epub 2012 Mar 5. PMID 22392168
- [Background] Corrigendum to "Analgesic Effect of Maternal Human Milk Odor on Premature Neonates: A Randomized Controlled Trial". J Hum Lact. 2017 Nov;33(4):822. doi: 10.1177/0890334417733738. PMID 28984527
- [Background] Badiee Z, Asghari M, Mohammadizadeh M. The calming effect of maternal breast milk odor on premature infants. Pediatr Neonatol. 2013 Oct;54(5):322-5. doi: 10.1016/j.pedneo.2013.04.004. Epub 2013 May 23. PMID 23707040
- [Background] Blass EM. Milk-induced hypoalgesia in human newborns. Pediatrics. 1997 Jun;99(6):825-9. doi: 10.1542/peds.99.6.825. PMID 9164777
- [Derived] Velumula PK, Elbakoush F, Tabb C 2nd, Farooqi A, Lulic-Botica M, Jani S, Natarajan G, Bajaj M. Breast milk vs 24% sucrose for procedural pain relief in preterm neonates: a non-inferiority randomized controlled trial. J Perinatol. 2022 Jul;42(7):914-919. doi: 10.1038/s41372-022-01352-2. Epub 2022 Feb 23. PMID 35197549